CLINICAL TRIAL: NCT02918448
Title: A Resistance Training Program Decreases the Risk of Metabolic Syndrome and Inflammatory Biomarkers in Older Adult Women: A Randomized Controlled Trial
Brief Title: Resistance Training and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Crisieli Maria Tomeleri, Doctor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UEL10656/2012
Record Dates: First submitted 2016-09-21; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taining group (Experimental): training group that performed the resistance program. All participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays. The RT program was performed in the following order: chest press, horizontal leg press, seated row, knee extension, preacher curl (free weights), leg curl, triceps pushdown, and seated calf raise. Participants of the TG performed 3 sets of 10-15 repetition maximums. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise
  Interventions: Other: Training group
- control group (No Intervention): control group that did not perform any type of physical exercise

INTERVENTIONS:
Other: Training group — The investigation was carried out over a period of 18 weeks, with 12 weeks dedicated to the RT program and 6 weeks allocated for measurements. Anthropometric, one repetition maximum tests (1RM), body composition, blood pressure (BP), dietary intake and blood sample measurements were performed in weeks 1-3, and 16-18. A supervised progressive RT program was performed between weeks 4-15 by the training group.
  Arms: Taining group

SUMMARY:
Metabolic syndrome (MetS) is a multicomponent disorder closely linked to low grade inflammation, and cardiovascular disease (CVD). The aim of this study was to investigate the effects of a 12-week resistance training (RT) program on body composition, risk factors for metabolic syndrome (MetS), and inflammatory biomarkers in older adult women

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of a 12-week resistance training (RT) program on body composition, risk factors for metabolic syndrome (MetS), and inflammatory biomarkers in older adult women. For the selection of the sample all participants completed a health history and we adopted the following inclusion criteria: 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction, not receiving hormonal replacement therapy, and not performing any regular physical exercise more than once a week in the six months preceding the beginning of the investigation. Participants passed a diagnostic graded exercise stress test with a 12-lead electrocardiogram, reviewed by a cardiologist, and were released with no restrictions for participation in this investigation. Written informed consent was obtained from all participants after being provided with a detailed description of investigation procedures. This investigation was conducted according to the Declaration of Helsinki and approved by the local University Ethics Committee. The investigation was carried out over a period of 18 weeks, with 12 weeks dedicated to the RT program and 6 weeks allocated for measurements. Anthropometric, one repetition maximum tests (1RM), body composition, blood pressure (BP), dietary intake and blood sample measurements were performed in weeks 1-3, and 16-18. It was also evaluated the Z-score risk for metabolic syndrome, which was based on the risk factors for metabolic syndrome. A supervised progressive RT program was performed between weeks 4-15 by the training group. The CG did not perform any type of physical exercise during this period. The RT training program was based on recommendations for RT in an older population. All participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays. The RT program was performed in the following order: chest press, horizontal leg press, seated row, knee extension, preacher curl (free weights), leg curl, triceps pushdown, and seated calf raise. Participants of the TG performed 3 sets of 10-15 repetition maximums. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise. Instructors adjusted the loads of each exercise according to the subject's ability and improvements in exercise capacity throughout the investigation in order to ensure that the subjects were exercising with as much resistance as possible while maintaining proper exercise technique.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction, not receiving hormonal replacement therapy, and not performing any regular physical exercise more than once a week in the six months preceding the beginning of the investigation.
* Participants passed a diagnostic graded exercise stress test with a 12-lead electrocardiogram, reviewed by a cardiologist, and were released with no restrictions for participation in this investigation.

Exclusion Criteria:

* All subjects not participating in 85% of the total sessions of training or withdrawl

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory Biomarkes | Baseline and 12 weeks
  Measurements of TNF-α, and IL-6, were determined by enzyme-linked immunosorbent assay (ELISA), according to the speciﬁcations of the manufacturer (Quantikine High Sensitivity Kit, R&D Systems, Minneapolis, MN) and performed in a microplate reader Perkin Elmer, model EnSpire (Waltham, MA, USA). The results are presented in picograms per milliliter (pg/ml). All samples were determined in duplicate to guarantee the precision of the results.
Change in Lipid and Glycemic Profiles | Baseline and 12 weeks
  Venous blood samples were collected after a 12 h fast and a minimum of 72 h after the final physical exercise session. Five milliliters were withdrawn from a prominent superficial vein in the antecubital space using a clean venous puncture with minimal stasis and placed in a tube containing ethylenediaminetetraacetic acid (EDTA) as an anticoagulant and conservant and a tube without coagulant. All samples were centrifuged for 15 min, and plasma or serum aliquots were stored at -80ºC until assayed. Measurements of glucose, high-density lipoprotein (HDL-C), and triglycerides (TG), were immediately determined in a specialized laboratory at University Hospital. The analyses were carried out using a biochemical auto-analyzer system (Dimension RxL Max - Siemens Dade Behring) according to established methods in the literature, consistent with the manufacturer's recommendations. The results are presented in milligrams per deciliter (mg/dL)
Change in Homeostasis Model Assessment (HOMA-IR) | Baseline and 12 weeks
  Insulin was measured by chemiluminescence using a Liaison XL analyzer (DiaSorin S.p.A., Saluggia, Italy). The homeostasis model assessment (HOMA-IR) was calculated by the formula: fasting insulin (μUI/ml) x fasting glucose (mmol/L)/22.5. Inter- and intra-assay coefficients of variation were <10% as determined in human plasma.
Change in Blood Pressure | Baseline and 12 weeks
  Resting BP assessment was performed using automatic oscillometric equipment (Omron HEM-742INT model, Omron Corporation, Kyoto, Kansai, Japan). Participants attended the laboratory on three different days and, during each visit, remained seated at rest for five minutes with the cuff of the equipment in place on the right arm. Subsequently, several BP measurements were performed at one-minute intervals in order to obtain three consecutive measurements where the difference in Systolic BP (SBP) and Diastolic BP (DBP) readings differed by no more than 4 mmHg. The median of the three measurements for each day was averaged across the three visits. Mean arterial pressure (MAP) was calculated using the formula MAP= DBP + 1/3 (SBP-DBP). The results are presented in (mmHg)
Change in Metabolic Syndrome Z score | Baseline and 12 weeks
  The metabolic syndrome Z score was also used in the present investigation as a continuous score of the five metabolic syndrome variables in agreement with the Adult Treatment Panel III criteria. A Z score was calculated for each variable using individual data, and standard deviations of data for the entire group at baseline (n = 53) and post intervention (n =47). The equation used to calculate the metabolic syndrome Z-score was Z score pre intervention = [(50 - HDL)/11.1 (11.9m2) + (TG - 150)/36.8 (42.1)] + [(fasting blood glucose - 100)/14.8 (13.7 m2)] + [(waist circumference - 88)/9.4 (9.9 m2)] + [(mean arterial pressure - 100)/6.4 (7.7) m2], and Z score post intervention= [(50 - HDL)/11.9 + (TG - 150)/42.1)] + [(fasting blood glucose - 100)/13.7)] + [(waist circumference - 88)/9.9] + [(mean arterial pressure - 100)/7.7)].
Change in C-reative Protein | Baseline and 12 weeks
  Measurements of serum levels of high-sensitivity CRP were carried out using a biochemical auto-analyzer system (Dimension RxL Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. The results are presented in milligram/liter (mg/L)
Change in Body Composition | Baseline and 12 weeks
  Whole-body dual-energy X-ray absorptiometry (DXA) scans (Lunar Prodigy, model NRL 41990, GE Lunar, Madison, WI) were used to assess body fat, trunk fat and appendicular lean soft tissue. The total skeletal muscle mass was estimated by the predictive equation proposed by Kim et al.. Prior to scanning, participants were instructed to remove all objects containing metal. Scans were performed with the subjects lying in the supine position along the table's longitudinal centerline axis. Feet were taped together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. Both calibration and analysis were carried out by a skilled laboratory technician. Equipment calibration followed the manufacturer's recommendations. The software generated standard lines that set apart the limbs from the trunk and head. These lines were adjusted by the same technician using specific anatomical points determined by the manufacturer.
Change in Waist Circumference | Baseline and 12 weeks
  Measures of waist circumference (WC) were obtained according to procedures established in the literature. The results are presented in centimeters (cm).

SECONDARY OUTCOMES:
Changes in Anthropometry Parameters | Baseline and 12 weeks
  Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale (Balmak, Laboratory Equipment Labstore, Curitiba, Paraná, Brazil), with the participants wearing light workout clothing and no shoes. Height was measured with a stadiometer attached to the scale to the nearest 0.1 cm, with subjects standing without shoes. Body mass index was calculated as body mass in kilograms divided by the square of height in meters.
Changes in Total Strength | Baseline and 12 weeks
  Maximal dynamic strength was evaluated using the 1RM test assessed in the chest press (CP), knee extension (KE), and preacher curl (PC) exercises, performed in this exact order. Testing for each exercise was preceded by a warm-up set (6-10 repetitions), with approximately 50% of the estimated load used in the first attempt of the 1RM. This warm-up was also used to familiarize the subjects with the testing equipment and lifting technique. The testing procedure was initiated 2 minutes after the warm-up. The subjects were instructed to try to accomplish two repetitions with the imposed load and were given three attempts in both exercises. The rest period was 3 to 5 min between each attempt, and 5 min between exercises. The 1RM was recorded as the final load lifted in which the subject was able to complete only one single maximal execution. Total strength was determined by the sum of the 3 exercises.
Changes in Dietary intake | Baseline and 12 weeks
  Participants were instructed by a dietitian to complete a food record on three nonconsecutive days (two week days and one weekend day) pre- and post-intervention. Participants were given specific instructions regarding the recording of portion sizes and quantities to identify all food and fluid intake, in addition to viewing food models in order to enhance precision. Total energy intake, protein, carbohydrate, and lipid content were calculated using nutrition analysis software (Avanutri Processor Nutrition Software, Rio de Janeiro, Brazil; Version 3.1.4).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Conceicao MS, Bonganha V, Vechin FC, Berton RP, Lixandrao ME, Nogueira FR, de Souza GV, Chacon-Mikahil MP, Libardi CA. Sixteen weeks of resistance training can decrease the risk of metabolic syndrome in healthy postmenopausal women. Clin Interv Aging. 2013;8:1221-8. doi: 10.2147/CIA.S44245. Epub 2013 Sep 16. PMID 24072967
- [Result] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Costa F; American Heart Association; National Heart, Lung, and Blood Institute. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute Scientific Statement. Circulation. 2005 Oct 25;112(17):2735-52. doi: 10.1161/CIRCULATIONAHA.105.169404. Epub 2005 Sep 12. No abstract available. PMID 16157765
- [Result] Kim J, Wang Z, Heymsfield SB, Baumgartner RN, Gallagher D. Total-body skeletal muscle mass: estimation by a new dual-energy X-ray absorptiometry method. Am J Clin Nutr. 2002 Aug;76(2):378-83. doi: 10.1093/ajcn/76.2.378. PMID 12145010